CLINICAL TRIAL: NCT03839771
Title: A Phase 3, Multicenter, Double-blind, Randomized, Placebo-controlled Study of Ivosidenib or Enasidenib in Combination With Induction Therapy and Consolidation Therapy Followed by Maintenance Therapy in Patients With Newly Diagnosed Acute Myeloid Leukemia or Myelodysplastic Syndrome With Excess Blasts-2, With an IDH1 or IDH2 Mutation, Respectively, Eligible for Intensive Chemotherapy.
Brief Title: A Study of Ivosidenib or Enasidenib in Combination With Induction Therapy and Consolidation Therapy, Followed by Maintenance Therapy in Patients With Newly Diagnosed Acute Myeloid Leukemia or Myedysplastic Syndrome EB2, With an IDH1 or IDH2 Mutation, Respectively, Eligible for Intensive Chemotherapy
Acronym: HOVON150AML
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Stichting Hemato-Oncologie voor Volwassenen Nederland (Other)
Collaborators: Deutsch-Österreichische Studiengruppe Akute Myeloische Leukämie (AMLSG) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HO150; 2018-000451-41 (EudraCT Number)
Record Dates: First submitted 2019-02-06; First posted 2019-02-15 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome With Excess Blasts-2
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — ivosidenib; enasidenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Placebo (Placebo Comparator): Cycle 1: day 1-start cycle 2 | Cycle 2: day 1 - start consolidation treatment | Consolidation treatment: day 1 - start maintenance | Maintenance treatment: day 1- day 730 (2 years) |
  The dosage for Placebo for AG-120 (IDH1): 500 mg dose/day
  The dosage for Placebo for AG-221 (IDH2): 100mg dose/day
  Interventions: Drug: Placebo for AG-120; Drug: Placebo for AG-221
- Arm B: Ivosidenib (IDH1) or Enasidenib (IDH2) (Experimental): Cycle 1: day 1-start cycle 2 | Cycle 2: day 1 - start consolidation treatment | Consolidation treatment: day 1 - start maintenance | Maintenance treatment: day 1- day 730 (2 years) |
  The dosage for AG-120 (IDH1): 500 mg dose/day
  The dosage for AG-221 (IDH2): 100mg dose/day
  Interventions: Drug: AG-120; Drug: AG-221

INTERVENTIONS:
Drug: AG-120 — 250mg tablets
  Other Names: Ivosidenib
  Arms: Arm B: Ivosidenib (IDH1) or Enasidenib (IDH2)
Drug: Placebo for AG-120 — 250mg tablets
  Arms: Arm A: Placebo
Drug: AG-221 — 100mg tablets
  Other Names: Enasidenib
  Arms: Arm B: Ivosidenib (IDH1) or Enasidenib (IDH2)
Drug: Placebo for AG-221 — 100mg tablets
  Arms: Arm A: Placebo

SUMMARY:
AML and MDS-EB2 are malignancies of the bone marrow. The standard treatment for these diseases is chemotherapy. Patients participating have a special type of this disease because the leukemia cells (blasts) have developed an error in the genetic material (DNA). This error is called an IDH1 mutation or an IDH2 mutation (a mutation is a change in the DNA), which leads to changes in specific substances in the leukemia cells. This trial will investigate whether the addition of the new drugs Ivosidenib (for patients with IDH1 mutation) or Enasidenib (for patients with IDH2 mutation) to the standard treatment of chemotherapy controle the disease more effectively and for a longer period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Newly diagnosed AML or MDS-EB2 defined according to WHO criteria, with a documented IDH1 or IDH2 gene mutation (as determined by the clinical trial assay) at a specific site (IDH1 R132, IDH2 R140, IDH2 R172). AML may be secondary to prior hematological disorders, including MDS, and/or therapy-related (in which prior disease should have been documented to have existed for at least 3 months). Patients may have had previous treatment with hypomethylating agents (HMAs) for MDS. HMAs have to be stopped at least four weeks before registration
* Patients with dual mutant FLT3 and IDH1 or IDH2 mutations may be enrolled only if, for medical or other reasons, treatment with a FLT3 inhibitor is not considered.
* Considered to be eligible for intensive chemotherapy.
* ECOG/WHO performance status ≤ 2
* Adequate hepatic function as evidenced by:

  * Serum total bilirubin ≤ 2.5 × upper limit of normal (ULN) unless considered due to Gilbert's disease (e.g. a mutation in UGT1A1) (only for patients in IDH2 cohort), or leukemic involvement of the liver - following written approval by the (Co)Principal Investigator.
  * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 3.0 × ULN, unless considered due to leukemic involvement of the liver, following written approval by the Principal Investigator.
* Adequate renal function as evidenced by creatinine clearance > 40 mL/min based on the Cockroft-Gault formula for glomerular filtration rate (GFR).
* Able to understand and willing to sign an informed consent form (ICF).
* Written informed consent

Female patient must either:

o Be of nonchildbearing potential: Postmenopausal (defined as at least 1 year without any menses) prior to screening, or Documented surgically sterile or status posthysterectomy (at least 1 month prior to screening)

o Or, if of childbearing potential: Agree not to try to become pregnant during the study and for 6 months after the final study drug administration And have a negative urine or serum pregnancy test at screening And, if heterosexually active, agree to consistently use highly effective* contraception per locally accepted standards in addition to a barrier method starting at screening and throughout the study period and for 6 months after the final study drug administration.

* Highly effective forms of birth control include:

  * Consistent and correct usage of established hormonal contraceptives that inhibit ovulation,
  * Established intrauterine device (IUD) or intrauterine system (IUS),
  * Bilateral tubal occlusion,
  * Vasectomy (A vasectomy is a highly effective contraception method provided the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used.)
  * Male is sterile due to a bilateral orchiectomy.
  * Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual activity during the entire period of risk associated with the study drug. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the patient.
* List is not all inclusive. Prior to enrollment, the investigator is responsible for confirming patient will utilize highly effective forms of birth control per the requirements of the CTFG Guidance document 'Recommendations related to contraception and pregnancy testing in clinical trials', September 2014 (and any updates thereof) during the protocol defined period.

  * Female patient must agree not to breastfeed starting at screening and throughout the study period, and for 2 months and 1 week after the final study drug administration.
  * Female patient must not donate ova starting at screening and throughout the study period, and for 6 months after the final study drug administration.

    * Male patient and their female partners who are of childbearing potential must be using highly effective contraception per locally accepted standards in addition to a barrier method starting at screening and continue throughout the study period and for 4 months and 1 week after the final study drug administration
    * Male patient must not donate sperm starting at screening and throughout the study period and for 4 months and 1 week after the final study drug administration.

      * Subject agrees not to participate in another interventional study while on treatment

Exclusion Criteria:

* Prior chemotherapy for AML or MDS-EB2 (with the exception of HMA). Hydroxyurea is allowed for the control of peripheral leukemic blasts in patients with leukocytosis (e.g., white blood cell [WBC] counts > 30x109/L).
* Dual IDH1 and IDH2 mutations.
* Acute promyelocytic leukemia (APL) with PML-RARA or one of the other pathognomonic variant fusion genes/chromosome translocations.
* Blast crisis after chronic myeloid leukemia (CML).
* Known allergy or suspected hypersensitivity to Ivosidenib or Enasidenib and/or any exipients.
* Taking medications with narrow therapeutic windows with potential interaction with investigational medication (see Appendix I), unless the patient can be transferred to other medications prior to enrolling or unless the medications can be properly monitored during the study.
* Taking P-glycoprotein (P-gp) or breast cancer resistance protein (BCRP) transporter-sensitive substrate medications (see Appendix J) unless the patient can be transferred to other medications within ≥ 5 half-lives prior to administration of ivosidenib or enasidenib, or unless the medications can be properly monitored during the study.
* Breast feeding at the start of study treatment.
* Active infection, including hepatitis B or C or HIV infection that is uncontrolled at randomization. An infection controlled with an approved or closely monitored antibiotic/antiviral/antifungal treatment is allowed.
* Patients with a currently active second malignancy. Patients are not considered to have a currently active malignancy if they have completed therapy and are considered by their physician to be at < 30% risk of relapse within one year. However, patients with the following history/concurrent conditions are allowed:

  * Basal or squamous cell carcinoma of the skin
  * Carcinoma in situ of the cervix
  * Carcinoma in situ of the breast
  * Incidental histologic finding of prostate cancer
* Significant active cardiac disease within 6 months prior to the start of study treatment, including New York Heart Association (NYHA) Class III or IV congestive heart failure (appendix G); myocardial infarction, unstable angina and/or stroke; or left ventricular ejection fraction (LVEF) < 40% by ultrasound or MUGA scan obtained within 28 days prior to the start of study treatment.
* QTc interval using Fridericia's formula (QTcF) ≥ 450 msec or other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure,family history of long QT interval syndrome). Prolonged QTc interval associated with bundle branch block or pacemaking is permitted with written approval of the Principal Investigator.
* Taking medications that are known to prolong the QT interval (see Appendix K), unless deemed critical and without a suitable alternative. In those cases, they may be administered, but with proper monitoring (see section 10.2, Table 13).
* Dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of orally administered drugs.
* Clinical symptoms suggestive of active central nervous system (CNS) leukemia or known CNS leukemia. Evaluation of cerebrospinal fluid (CSF) during screening is only required if there is a clinical suspicion of CNS involvement by leukemia during screening.
* A known medical history of progressive multifocal leukoencephalopathy (PML).
* Immediately life-threatening, severe complications of leukemia such as uncontrolled bleeding, pneumonia with hypoxia or shock, and/or severe disseminated intravascular coagulation
* Any other medical condition deemed by the Investigator to be likely to interfere with a patient's ability to give informed consent or participate in the study.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 968 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2027-04-17 (Estimated); Study Completion 2034-09-19 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | Approximately up to 60 months following first patient enrollment
  EFS is defined as the time from randomization to failure to achieve CR or CRi after remission induction, death after achieving CR or CRi or relapse after achieving CR or CRi, whichever occurs first. A patient is said to have failed to achieve CR or CRi after induction therapy, if his/her best response during or at completion of the induction treatment is less than CRi. Patients who achieved CR/CRi after remission induction and are not known to have relapsed or died will be censored at the date of last clinical assessment.

SECONDARY OUTCOMES:
Overall survival (OS) | Approximately up to 84 months following first patient enrollment
  OS is defined as the time from date of randomization to date of death due to any cause. Patients still alive or lost to follow up will be censored at the time they were last known to be alive.
Relapse-free survival (RFS) after CR/CRi | Approximately up to 60 months following first patient enrollment
  RFS is defined as time from the date of achievement of CR/CRi until relapse or death from any cause, whichever comes first. Patients still in first CR/CRi and alive or lost to follow up will be censored at the date of last clinical assessment.
Cumulative incidence of relapse (CIR) after CR/CRi | Approximately up to 60 months following first patient enrollment
  CIR is measured from the date of achievement of CR/CRi until the date of relapse. Patients not known to have relapsed will be censored on the date of last clinical assessment. Patients who died without relapse will be counted as a competing cause of failure.
Cumulative incidence of death (CID) after CR/CRi | Approximately up to 60 months following first patient enrollment
  CID is measured from the date of achievement of CR/CRi until the date of death from any cause. Patients not known to have died will be censored on the date they were last known to be alive. Patients who experienced relapse in CR/CRi will be counted as competing cause of failure.
Complete remission without minimal residual disease (CRMRD-) rate after induction cycle 2 | Approximately up to 60 months following first patient enrollment
  CRMRD- rate is defined as the percentage of patients who achieved CR or CRi with no evidence of MRD in bone marrow
Frequency and severity of adverse events according to CTCAE version 5.0 | Continuously throughout the study, starting from informed consent until 30 days following the last administration of any study drug
  Adverse events will be evaluated using the National Cancer Institute's Common Terminology Criteria for AEs (CTCAE) version 5.0
CR/CRi rates after induction cycle 1 and 2 | Approximately up to 60 months following first patient enrollment
  CR and CRi are determined by the Investigator based on the European LeukemiaNet (ELN2017) recommended response criteria
CR/CRi rate after remission induction (i.e., CR or CRi as best response during or at completion of induction therapy) | Approximately up to 60 months following first patient enrollment
  CR+CRi rate after remission induction is defined as the percentage of patients with best response of CR or CRi during or at completion of induction therapy
Time to hematopoietic recovery after each chemotherapy treatment cycle | Approximately up to 60 months following first patient enrollment
  Time to hematopoietic recovery is defined as the time from the start of the cycle until recovery
EQ-5D-5L visual analogue scale (VAS) | At entry, 1st day of maintenance, every 3 months during the first year of maintenance, every 6 months during the second year of maintenance until relapse or treatment discontinuation (approximately up to 84 months following first patient enrollment)
  The EQ-5D-5L is a 5 item questionnaire that assesses 5 domains including mobility, self-care, usual activities, pain/discomfort and anxiety/depression plus a visual analog scale rating "health today". Each domain has 5 levels. Each level has a 1 digit number expressing the level selected for that dimension. These levels are summed up and the self-rated health is recorded on a 20 cm vertical, visual analogue scale, with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'.
EORTC-QLQ-C30 global health status/QoL scale. | At entry, 1st day of maintenance, every 3 months during the first year of maintenance, every 6 months during the second year of maintenance until relapse or treatment discontinuation (approximately up to 84 months following first patient enrollment)
  The EORTC QLQ-C30 is a 30-item questionnaire that assesses 5 functional subdomains (physical functioning, role functioning, emotional functioning, cognitive functioning and social functioning), 1 global health status, 3 symptom subdomains (fatigue, nausea and vomiting and pain) and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Estimate the average of the items that contribute to the scale; this is the raw score. a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: B.J. Wouters, Principal Investigator — Erasmus MC / HOVON
Locations (181):
- Australia (21):
  - AU-Adelaide-FLINDERS, Adelaide
  - AU-Adelaide-RAH, Adelaide
  - AU-Brisbane-PAH, Brisbane
  - AU-Camperdown-RPA, Camperdown
  - AU-Canberra-CANBERRAHOSPITAL, Canberra
  - AU-Douglas-TOWNSVILLE, Douglas
  - AU-Hobart TAS-RHOBART, Hobart
  - AU-Launceston TAS-LAUNCESTON, Launceston
  - AU-Melbourne-ALFRED, Melbourne
  - AU-Melbourne-AUSTIN, Melbourne
  - AU-Melbourne-MONASH, Melbourne
  - AU-Melbourne-RMELBOURNE, Melbourne
  - AU-Melbourne-SVHM, Melbourne
  - AU-Perth-FSH, Perth
  - AU-Perth-RPH, Perth
  - AU-Perth-SCGH, Perth
  - AU-Sydney-CONCORD, Sydney
  - AU-Sydney-RNSH, Sydney
  - AU-Sydney-SVHS, Sydney
  - AU-Sydney-WSAH, Sydney
  - AU-Waratah-CALVARYMATER, Waratah
- Austria (4):
  - AT-Graz-MEDUNIGRAZ, Graz
  - AT-Innsbruck-IMED, Innsbruck
  - AT-Linz-ORDENSKLINIKUM, Linz
  - AT-Vienna-HANUSCH, Vienna
- Belgium (13):
  - BE-Antwerpen-ZNASTUIVENBERG, Antwerp
  - BE-Brugge-AZBRUGGE, Bruges
  - BE-Brussel-BORDET, Brussels
  - BE-Brussel-UZBRUSSEL, Brussels
  - BE-Bruxelles-STLUC, Brussels
  - BE-Gent-UZGENT, Ghent
  - BE-Haine-Saint-Paul-JOLIMONT, Haine-Saint-Paul
  - BE-Hasselt-VIRGAJESSE, Hasselt
  - BE-Leuven-UZLEUVEN, Leuven
  - BE-Liege-CHRCITADELLE, Liège
  - BE-Liege-CHULIEGE, Liège
  - BE-Roeselare-AZDELTA, Roeselare
  - BE-Yvoir-MONTGODINNE, Yvoir
- EE-Tartu-TARTU, Tartu, Estonia
- Finland (2):
  - FI-Helsinki-HUS, Helsinki
  - FI-Tampere-TAYS, Tampere
- France (37):
  - FR-Amiens-CHUAMIENS, Amiens
  - FR-Angers-CHUANGERS, Angers
  - FR-Argenteuil-CHARGENTEUIL, Argenteuil
  - FR-Bayonne-CHCOTEBASQUE, Bayonne
  - FR-Besançon Cedex-JEANMINJOZ, Besançon
  - FR-Bobigny-AVICENNE, Bobigny
  - FR-Chambery-CHMETROPOLESAVOIE, Chambéry
  - FR-Le Chesnay cedex-CHVERSAILLES, Chesnay
  - FR-Clamart-HIAPERCY, Clamart
  - FR-Clermont-Ferrand-ESTAING, Clermont-Ferrand
  - FR-Créteil cedex-CHUMONDOR, Créteil
  - FR-Grenoble cedex 9-CHUGRENOBLE, Grenoble
  - FR-Lens-CHLENS, Lens
  - FR-Lille-CHULILLE, Lille
  - FR-Limoges-CHULIMOGES, Limoges
  - FR-Lyon Pierre Benite cedex-LYONSUD, Lyon
  - FR-Lyon-LEONBERARD, Lyon
  - FR-Marseille-IPC, Marseille
  - FR-Montpellier-STELOI, Montpellier
  - FR-Mulhouse-GHRMSA, Mulhouse
  - FR-Nantes-CHUNANTES, Nantes
  - FR-Nice-CAL, Nice
  - FR-Nice-LARCHET, Nice
  - FR-Orléans-CHORLEANS, Orléans
  - FR-Paris cedex 10-SAINTLOUIS, Paris
  - FR-Paris cedex 12-SAINTANTOINE, Paris
  - FR-Paris cedex 15-NECKER, Paris
  - FR-Pessac Cedex-CHUBORDEAUX, Pessac
  - FR-Poitiers-CHUPOITERS, Poitiers
  - FR-Reims-CHREIMS, Reims
  - FR-Rennes cedex 9-CHURENNES, Rennes
  - FR-Rouen cedex-BECQUEREL, Rouen
  - FR-Strasbourg cedex-HAUTEPIERRE, Strasbourg
  - FR-Toulouse-CHUTOULOUSE, Toulouse
  - FR-Tours cedex-BRETONNEAU, Tours
  - FR-Vandoeuvre Les Nancy-CHRUNANCY, Vandœuvre-lès-Nancy
  - FR-Villejuif-GUSTAVEROUSSY, Villejuif
- Germany (48):
  - DE-Bad Saarow-HELIOSBADSAAROW, Bad Saarow
  - DE-Berlin-CAMPUSBENFRANKLIN, Berlin
  - DE-Berlin-CAMPUSVIRCHOW, Berlin
  - DE-Berlin-VIVANTESNEUKOLLN, Berlin
  - DE-Berlin-VIVANTESURBAN, Berlin
  - DE-Bochum-RUB, Bochum
  - DE-Bonn-UNIBONN, Bonn
  - DE-Braunschweig-KLINIKUMBRAUNSCHWEIG, Braunschweig
  - DE-Bremen-KBM, Bremen
  - DE-Dortmund-JOHODORTMUND, Dortmund
  - DE-Düsseldorf-MEDUNIDUESSELDORF, Düsseldorf
  - DE-Essen-KEM, Essen
  - DE-Esslingen-KLINIKUMESSLINGEN, Esslingen am Neckar
  - DE-Flensburg-MALTESER, Flensburg
  - DE-Giessen-UKGM, Giessen
  - DE-Goch-KKLE, Goch
  - DE-Hamburg-ASKLEPIOSSTGEORG, Hamburg
  - DE-Hamburg-ASKLEPIOS, Hamburg
  - DE-Hamburg-UKE, Hamburg
  - DE-Hamm-EVKHAMM, Hamm
  - DE-Hanau-KLINIKUMHANAU, Hanau
  - DE-Hannover-MHHANNOVER, Hanover
  - DE-Hannover-SILOAHKRH, Hanover
  - DE-Herne-MARIENHOSPITALHERNE, Herne
  - DE-Homburg-UNIKLINIKSAARLAND, Homburg
  - DE-Karlsruhe-KLINIKUMKARLSRUHE, Karlsruhe
  - DE-Lebach-CARITASKHLEBACH, Lebach
  - DE-Lemgo-KLINIKUMLIPPE, Lemgo
  - DE-Ludwigshafen-KLILU, Ludwigshafen
  - DE-Luedenscheid-KLINIKUMLUEDENSCHEID, Lüdenscheid
  - DE-Magdeburg-OVGU, Magdeburg
  - DE-Mainz-KLINKUNIMAINZ, Mainz
  - DE-Mainz-UNIMEDIZINMAINZ, Mainz
  - DE-Meschede-HOCHSAUERLAND, Meschede
  - DE-Minden-MUEHLENKREISKLINKEN, Minden
  - DE-München-IRZTUM, München
  - DE-München-MEDUNIMUNCHIN, München
  - DE-Offenburg-ORTENAUKLINIKUM, Offenburg
  - DE-Oldenburg-KLINIKUMOLDENBURG, Oldenburg
  - DE-Passau-KLINIKUMPASSAU, Passau
  - DE-Stuttgart-DIAKSTUTTGART, Stuttgart
  - DE-Stuttgart-KLINIKUMSTUTTGART, Stuttgart
  - DE-Traunstein-TSSOB, Traunstein
  - DE-Trier-MUTTERHAUS, Trier
  - DE-Tübingen-MEDUNITUEBINGEN, Tübingen
  - DE-Ulm-UNIKLINKULM, Ulm
  - DE-Villingen-Schwenningen-SBKVS, Villingen-Schwenningen
  - DE-Wuppertal-HELIOSGESUNDHEIT, Wuppertal
- Ireland (4):
  - IE-Cork-CUH, Cork
  - IE-Dublin 8-STJAMES, Dublin
  - IE-Dublin 9-BEAUMONT, Dublin
  - IE-Galway-UHGALWAY, Galway
- LT-Vilnius-SANTA, Vilnius, Lithuania
- LU-Luxembourg-CHL, Luxembourg, Luxembourg
- Netherlands (21):
  - NL-Den Bosch-JBZ, 's-Hertogenbosch
  - NL-Amersfoort-MEANDERMC, Amersfoort
  - NL-Amsterdam-AMC, Amsterdam
  - NL-Amsterdam-OLVG, Amsterdam
  - NL-Amsterdam-VUMC, Amsterdam
  - NL-Arnhem-RIJNSTATE, Arnhem
  - NL-Breda-AMPHIA, Breda
  - NL-Delft-RDGG, Delft
  - NL-Dordrecht-ASZ, Dordrecht
  - NL-Eindhoven-MAXIMAMC, Eindhoven
  - NL-Enschede-MST, Enschede
  - NL-Groningen-UMCG, Groningen
  - NL-Leeuwarden-MCL, Leeuwarden
  - NL-Leiden-LUMC, Leiden
  - NL-Maastricht-MUMC, Maastricht
  - NL-Nieuwegein-ANTONIUS, Nieuwegein
  - NL-Nijmegen-RADBOUDUMC, Nijmegen
  - NL-Rotterdam-ErasmusMC, Rotterdam
  - NL-Den Haag-HAGA, The Hague
  - NL-Utrecht-UMCUTRECHT, Utrecht
  - NL-Zwolle-ISALA, Zwolle
- Norway (5):
  - NO-Bergen-HELSEBERGEN, Bergen
  - NO-Oslo-OSLOUH, Oslo
  - NO-Stavanger-HELSESTAVANGER, Stavanger
  - NO-Tromsø-NORTHNOORWEGEN, Tromsø
  - NO-Trondheim-STOLAV, Trondheim
- Spain (12):
  - ES-Barcelona-CLINICUB, Barcelona
  - ES-Barcelona-GERMANTRIALS, Barcelona
  - ES-Barcelona-ICODURANREYNALS, Barcelona
  - ES-Barcelona-MUTUATERRASSA, Barcelona
  - ES-Barcelona-PARCDESALUTMAR, Barcelona
  - ES-Barcelona-SANTPAU, Barcelona
  - ES-Barcelona-VHEBRON, Barcelona
  - ES-Girona-ICSTRUETA, Girona
  - ES-Madrid-CSGREGORIOMARANON, Madrid
  - ES-Palma-SSIB, Palma
  - ES-Tarragona-JOAN, Tarragona
  - ES-Valencia-MALVARROSA, Valencia
- Sweden (3):
  - SE-Lund-SUH, Lund
  - SE-Stockholm-KAROLINSKAHUDDINGE, Stockholm
  - SE-Uppsala-UPPSALAUH, Uppsala
- Switzerland (8):
  - CH-Basel-USB, Basel
  - CH-Bellinzona-IOSI, Bellinzona
  - CH-Bern-INSEL, Bern
  - CH-Fribourg-HFR, Fribourg
  - CH-Geneve (14)-HCUGE, Geneva
  - CH-Luzern-LUKS, Lucerne
  - CH-St. Gallen-KSSG, Sankt Gallen
  - CH-Zürich-USZ, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: HOVON website — http://www.hovon.nl